CLINICAL TRIAL: NCT00115427
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial of Liatermin (r-metHuGDNF) Administered by Bilateral Intraputaminal (IPu) Infusion to Subjects With Idiopathic Parkinson's Disease
Brief Title: Study of Liatermin (r-metHuGDNF) Administered by Bilateral Intraputaminal (IPu) Infusion to Subjects With Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020168
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Bilateral, Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Glial Cell Line-Derived Neurotrophic Factor

INTERVENTIONS:
Drug: Liatermin (r-metHuGDNF)

SUMMARY:
This randomized study was designed to evaluate the efficacy and safety of IPu-infused liatermin (15mg/putamen/day) compared with placebo in subjects with symptomatic, levodopa-response Parkinson's disease. This study consisted of a 90-day evaluation period followed by implantation of the IPu delivery system and then a 6-month double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of bilateral, idiopathic Parkinson's disease

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03

PRIMARY OUTCOMES:
United Parkinson's Disease Rating Scale

SECONDARY OUTCOMES:
Timed Motor Tests
Dyskinesia ratings
Diary ratings
Patient reported outcomes measures

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20020168.pdf